CLINICAL TRIAL: NCT05466942
Title: RDS MultiSense® SpO2 Calibration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhythm Diagnostic Systems (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR 2022-465
Record Dates: First submitted 2022-07-08; First posted 2022-07-20 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Hypoxia
Keywords: Hypoxia; Pulse Oximetry; SpO2; Remote monitoring; Connected device; Real-time monitoring
MeSH Terms: conditions — Hypoxia | interventions — Respiratory Rate; Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Controled Hypoxia - Healthy volunteer (Other): Male and female subjects, ranging in pigmentation from light to dark
  Interventions: Device: Pulse Oximeter, Respiratory Rate, Heart Rate

INTERVENTIONS:
Device: Pulse Oximeter, Respiratory Rate, Heart Rate — Measurement of physiological parameters

SUMMARY:
Data will be collected with the MultiSense® pulse oximetry system during non-motion conditions over the range of 70-100%. A Clinimark reference system, previously correlated to arterial blood CO-Oximetry will be the basis for comparison. A minimum of fifteen (15) up to fifty (50) healthy adult subjects, ranging in pigmentation from light to dark, with at least six (6) subjects with dark pigmentation (Fitzpatrick 5-6), will be enrolled in the study to meet the study design requirements defined by ISO 80601-2-61 and by the FDA's Guidance for Pulse Oximeters (March 4, 2013). SpO2 data will be evaluated during non-motion conditions. SpO2 data will be evaluated during stable step plateaus of induced hypoxic levels. The investigational device will be placed on the thorax of the subjects (patch on the upper back and external electrode on the right pectoral). Simultaneous data collection will be set up for the reference and the systems under test.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have the ability to understand and provide written informed consent
* Subject is 18 to 50 years of age
* Subject must be willing and able to comply with study procedures and duration
* Subject is a non-smoker or who has not smoked within 2 days prior to the study.
* Male or female of any race
* Subject demographics include a range of skin pigmentations, including at least 3 darkly pigmented subjects or 15% of the subject pool, whichever is larger.

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Compromised circulation, injury, or physical malformation of fingers, toes, hands, ears or forehead/skull or other sensor sites, tattoo in the optical path which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
* Females who are pregnant, who are trying to get pregnant, (confirmed by positive urine pregnancy test unless the subject is known to be not of child-bearing potential)
* Subjects who have smoked in the last 2 days with COHb levels >3% as assessed with a Masimo Radical 7 (Rainbow)
* Subjects with known respiratory conditions (self-reported)
* Subjects with known heart or cardiovascular conditions (self-reported, except for blood pressure and ECG review) or with an implantable active medical device such as pacemaker or automatic defibrillator
* Self-reported health conditions as identified in the Health Assessment Form (self-reported)
* Subjects with severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors (self-reported)
* Unwillingness or inability to remove colored nail polish from test digits.
* Unwillingness to have chest or other test site shaved
* Other known health condition, should be considered upon disclosure in health assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Determination of the quality of measurements of arterial blood saturation (SpO2) provided by the MultiSense® system in comparison to measurements made with a reference Pulse Oximetry System, in terms of accuracy. | from device placement to device removal, assessed up to 3 hours
  Accuracy is defined as an average measurement variation less than 3.5% of the mean value to the reference standard. Reference Pulse Oximetry Systems, previously compared to Reference CO-Oximetry will be used as the basis for comparison. The study population will include 15 to 50 subjects. The data for analysis will be equally distributed across the range of 70-100%. All data will be used for the analysis unless identified as unstable by the control oximeter. Data that is found to be unstable will be removed prior to the comparative analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinimark LLC, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No